CLINICAL TRIAL: NCT04166071
Title: Revisiting Safety Signals: Examining a Separate Safety Mechanism for Social Support Figures
Brief Title: Opioids and Social Support Enhanced Extinction Effects
Acronym: SSO
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Naomi Eisenberger, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: SSO
Record Dates: First submitted 2019-11-05; First posted 2019-11-18 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Fear
Keywords: social support; fear extinction
MeSH Terms: interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Naltrexone (Active Comparator)
  Interventions: Drug: Naltrexone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone — Half of the participants will be randomly assigned to take one dose of naltrexone (50mg, capsule form) during the experimental session
  Arms: Naltrexone
Drug: Placebo — Half of the participants will be randomly assigned to take a placebo capsule during the experimental session
  Arms: Placebo

SUMMARY:
University of California, Los Angeles researchers will recruit healthy participants (age 18-35) to participate in a study examining whether the administration of naltrexone, an opioid antagonist, eliminates the ability of social support figure reminders to enhance fear extinction--a process during which a threatening cue is learned to not predict a negative or threatening outcome (i.e., electric shock) by being repeatedly presented in the absence of that outcome.

After undergoing an email screening, a telephone screening, an in lab screening, and a health screening, 60 participants will be enrolled in the study. During the experiment, 30 participants will be administered naltrexone and 30 participants will be administered placebo (both participants and experimenters will be blind to condition) before undergoing a fear extinction procedure in which threatening cues--cues that predict electric shock--will be paired with either an image of a social support figure (provided by participants) or a second threatening cue. These pairings will be presented repeatedly in the absence of shock in order for fear extinction to occur. Participants will return for a follow-up test to determine if fear extinction was successful.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults 18 and 35
* fluent in English
* no history of mental illness (including anxiety, depression, phobia, or any other mental health related disorder diagnosed by a mental health professional)

Exclusion Criteria:

* pregnant or planning to become pregnant during the experiment period
* presence of chronic mental illness (as determined by the report of a past diagnosis of mental illness by a physician or psychologist and/or the prescription of medication related to mental health disorder; including anxiety, depression, phobia, or any other diagnosed psychological disorder)
* chronic physical illness (as determined by past diagnosis and/or treatment by a physician)
* history of liver disease or abnormal liver function
* current and regular use of prescription medications related to mental health disorders or liver function
* previous history of fainting during blood draws
* difficulty or discomfort swallowing pills
* history of substance abuse or addiction (especially alcohol or opiate abuse)

Other exclusion criteria may apply.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Fear Response directly post-extinction | Directly following a fear extinction procedure (during the experiment session).
  presence of fear response as indicated by significantly higher galvanic skin response (GSR: an index of peripheral stress responding) to a previously learned fearful image (CS+) compared to a baseline comparator (CS-: never learned to be fearful).
Fear Response 24-hours post-extinction | 24 hours following the completion of the fear extinction procedure (during a follow-up fear reinstatement session).
  presence of fear response as indicated by significantly higher galvanic skin response (GSR: an index of peripheral stress responding) to a previously learned fearful image (CS+) compared to a baseline comparator (CS-: never learned to be fearful).

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Eisenberger, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - UCLA Department of Psychology, 5514 Pritzker Hall, Los Angeles, California
  - UCLA, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No